CLINICAL TRIAL: NCT01687881
Title: Is Chiropractic Spinal Manipulative Therapy an Efficient Treatment Option in Cervicogenic Headache? A Randomized Controlled Clinical Trial.
Brief Title: Is Chiropractic Spinal Manipulative Therapy an Efficient Treatment Option in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Chiropractic Association (Unknown)
Responsible Party: Principal Investigator, Aleksander Chaibi, PhD student, University Hospital, Akershus
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CEH-K34KSF-AHUS; 2829002 (Other: Research Centre, Akershus University Hospital)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cervicogenic Headache
Keywords: Chiropractic; Manipulative therapy; Cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham Chiropractic (Sham Comparator): Sham Chiropractic manipulative therapy.
  Interventions: Other: Sham Chiropractic
- Control group (No Intervention): No intervention: Control group.
- Chiropractic Spinal Manipulative Therapy (Active Comparator): Active intervention: Chiropractic Spinal Manipulative Therapy
  Interventions: Other: Chiropractic

INTERVENTIONS:
Other: Chiropractic — Chiropractic Spinal Manipulative Therapy
  Arms: Chiropractic Spinal Manipulative Therapy
Other: Sham Chiropractic — Sham manipulation
  Arms: Sham Chiropractic

SUMMARY:
This study will highlight and validate chiropractic spinal manipulative therapy (CSMT) for cervicogenic headache (CEH). If the method proves to be effective, it will provide a new non-pharmacological treatment option for CEH. This is especially important since pharmacological management has minor effect in CEH, and alternative treatment options are warranted. The applied methodology of the study will aim towards the highest possible research standards. This international study is a collaboration between Akershus University Hospital, Innlandet Hospital and University of Oslo (UiO), Norway and Macquarie University, Australia. The multidisciplinary professional backgrounds are physiotherapy, chiropractic and medicine. By increasing the methodological quality of the investigators research to a very high level, the investigators see the method to work as a guide to increase the quality of chiropractic research in the future, as previous randomized clinical trials (RCTs) of CEH used methodology showing room for improvement.

Study hypothesis:

CSMT using the Gonstead method reduces days with CEH by at least 25% as compared to placebo (sham manipulation, i.e. broad non-specific contact, non-directional, low velocity and low amplitude) and no intervention (control group).

DETAILED DESCRIPTION:
Cervicogenic headache (CEH) is a symptomatic headache characterized by chronic unilateral headache and symptoms and signs of neck involvement. CEH is often worsened by neck movement, sustained awkward head position, external pressure over the upper cervical or occipital region on the symptomatic side. Abolition of the headache following diagnostic anesthetic blocks of cervical structures or local factors in neck give evidence that the pain is attributed to a neck disorder or lesion. The prevalence of CEH is 0.2% in the general population of Akershus County, i.e. 9,000 Norwegians have CEH. However, the prevalence varies between 0.4-4.1% in studies applying less rigorous diagnostic criteria. The efficacy of pharmacological management in CEH is poor. Patients suffering from CEH are commonly treated with CSMT, but the methodology has one or more shortcomings in all studies. In addition, the RCTs mostly included participant with infrequent CEH and did not follow the recommended clinical guidelines by the International Headache Society (IHS) of intervention of at least three months. An analysis of the literature as well as a recent pilot study suggests that CSMT has an effect on headache intensity and duration, and medication intake. However, a randomized controlled clinical trial with high methodological quality on CEH still remains to be conducted.

The RCT is single blinded, placebo-controlled trial of CSMT using the Gonstead method vs. sham manipulation and control group. If the treatment shows to be effective, the participants whom receive sham manipulation or control will be offered true intervention after the follow-up period and free of charge. This study will follow the recommendations set by the clinical trial guidelines from the IHS, while the methodological quality control will in general follow previous suggested criteria and the CONSORT statements.

Patients will be recruited through Akershus University Hospital and Innlandet Hospital, Norway as well as through media advertising in Akershus and Oslo County. The diagnose is set by a chiropractor and a neurologist with experience in headache.

The clinical trials consist of three stages: Run-in, intervention (treatment) and follow-up.

One month of base line data collection where participants will fill-in a diagnostic headache diary. Baseline demographics and clinical characteristics will be presented in tables with mean and standard deviation (SD) for each group.

The participants will be randomized by drawing prepared sealed lots. Each lot includes three different interventions, i.e active treatment, sham manipulation and control group. The first three participants will draw from the same lot until all three interventions are used. The next lot with three interventions is then followed by the next three participants.

The RCTs will be conducted by an experienced chiropractor. Active treatment consists of CSMT using the Gonstead method. A specific contact, high velocity, low amplitude, short lever, with no recoil post adjustment directed to spinal biomechanical dysfunction diagnosed by standard chiropractic tests.

Follow-up at 3, 6 and 12 months post-treatment. During this period participants continue to fill in a diagnostic headache diary. The control group will also be included in this phase of the study.

The data will be analyzed with SPSS using standard statistical techniques.

The investigators based our calculation of sample size on migraine days from recent group comparison studies of topiramate (38). The investigators calculated that a sample size of 16 patients was required to detect a difference in mean reduction in monthly headache days of 2.5 with 80% power, with p=0.05 as level of significance, and assuming a common SD of 2.5 for active treatment and broad-based treatment groups.

Insurance is through "The Norwegian System of Compensation to Patients" (NPE) which is an independent national body, set up to process compensation claims from patients who have suffered an injury as a result of treatment under the Norwegian health service.

The Regional Committee for Medical Research Ethics (REK) in Norway and Norwegian Social Science Data Services approved the full PhD research protocol. The declaration of Helsinski is followed.

ELIGIBILITY:
Inclusion Criteria:

* CEH according to at least three major criteria of the CHISG not including occipital nerve blockage
* Age 18-70 years

Exclusion Criteria:

* Contraindication to spinal manipulation
* Chiropractic treatment within the last 12 months
* Radiculopathy
* Depression
* Pregnancy
* Participants whom become pregnant during the migraine trial will also be excluded from analysis from the time of pregnancy
* Participants who change their prophylactic medical regime for headaches will be excluded in the analysis from the time of change

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of headache days | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in number of headache days between active treatment and sham.
  2. 25% reduction in number of headache days between active treatment and control group.

SECONDARY OUTCOMES:
Headache duration | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in headache duration in hours between active treatment and sham.
  2. 25% reduction in headache duration in hours between active treatment and control group.
Self reported VAS | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% self-reported improvement on VAS between active treatment and sham.
  2. 25% self-reported improvement on VAS between active treatment and control group.
Headache index | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in headache index (frequency x duration x intensity) between active treatment and sham.
  2. 25% reduction in headache index between active treatment and control group.
Headache medication | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 50% reduction in headache medication between active treatment and sham.
  2. 50% reduction in headache medication between active treatment and control group.

OTHER OUTCOMES:
Sub-analysis on x-ray findings | Change formbaseline to post-treatment, 3, 6, 12 months follow-up
  Sub-analysis will be done on participants with structural deformities vs. normal x-ray findings.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Russell, Professor, Study Director — Head and Neck research Group, Research Centre, Akershus University Hospital
Locations (1):
- Research Centre, Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Background] Chaibi A, Russell MB. Manual therapies for cervicogenic headache: a systematic review. J Headache Pain. 2012 Jul;13(5):351-9. doi: 10.1007/s10194-012-0436-7. Epub 2012 Mar 30. PMID 22460941
- [Background] Chaibi A, Benth JS, Tuchin PJ, Russell MB. Chiropractic spinal manipulative therapy for cervicogenic headache: a study protocol of a single-blinded placebo-controlled randomized clinical trial. Springerplus. 2015 Dec 16;4:779. doi: 10.1186/s40064-015-1567-5. eCollection 2015. PMID 26697289
- [Result] Chaibi A, Knackstedt H, Tuchin PJ, Russell MB. Chiropractic spinal manipulative therapy for cervicogenic headache: a single-blinded, placebo, randomized controlled trial. BMC Res Notes. 2017 Jul 24;10(1):310. doi: 10.1186/s13104-017-2651-4. PMID 28738895